CLINICAL TRIAL: NCT06025357
Title: Effects of L-Citrulline Supplementation on Vascular Function During Fasted and Acute Hyperglycemia in Middle-aged and Older Women With Metabolic Syndrome
Brief Title: Effects of L-citrulline Supplementation on Vascular Function in Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Responsible Party: Principal Investigator, Arturo Figueroa, Arturo Figueroa, Principal Investigator, Texas Tech University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB2022-362
Record Dates: First submitted 2023-07-27; First posted 2023-09-06 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2023-08

CONDITIONS: Metabolic Syndrome; Menopause
Keywords: Endothelial function; Aortic Hemodynamics; Blood pressure; Obesity; Hypertension
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Hypertension

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Double (Participant, Investigator) Randomized, double-blind, placebo-controlled, parallel study design
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- L-citrulline (Experimental): L-citrulline: 10 grams/day
  Interventions: Dietary Supplement: L-Citrulline supplementation
- Placebo (Experimental): Microcrystalline Cellulose
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: L-Citrulline supplementation — 4 weeks of L-Citrulline supplementation (10 grams/day).
  Arms: L-citrulline
Dietary Supplement: Placebo — 4 weeks of microcrystalline Cellulose supplementation.
  Arms: Placebo

SUMMARY:
The objective of this project is to provide evidence that L-Citrulline (CIT) supplementation can improve vascular function in the fasted and acute hyperglycemia conditions in middle-aged and older women with metabolic syndrome.

DETAILED DESCRIPTION:
Using a double-blind, randomized, placebo-controlled, and parallel design, middle-aged and older women with metabolic syndrome will be randomized into receiving either CIT supplementation (10g/day) or placebo (Microcrystalline Cellulose) for 4 weeks.

The first visit will be approximately 1hr and 30 minutes. The 2nd and 3rd visits will each be approximately 2hrs and 30 minutes, separated by 4 weeks in between each visit. During visits 2 and 3, vascular measurements will be assessed in the fasted state and 30, 60, and 90 minutes after acute glucose ingestion (75g).

ELIGIBILITY:
Inclusion Criteria:

Must present at least 3 of the following 5 cardiometabolic risk factors

* Waist circumference ≥88 cm
* Fasting glucose between 100-125 mg/dL or HbA1c between 5.7-6.4%.
* Blood pressure ≥130 mm Hg
* Triglyceride ≥ 150 mg/dL
* HDL <50 mg/dL

The following are also inclusion criteria's:

* Women aged 45-79 years old
* Body mass index ≤ 39.9 kg/m2
* Sedentary (defined as < 120 min/week of exercise)
* Abstain from any dietary supplements with vascular effects for one month prior to the beginning of the study and until participation in study has terminated.

Exclusion Criteria:

* < 45 and > 79 years of age
* Use of medications and/or any supplements that may affect outcome variables (such as arginine-containing supplements, nitroglycerin, statin drugs, biguanides, insulin, beta blockers, statins, verapamil)
* Systolic blood pressure ≥ 160 mmHg
* BMI > 40 kg/m2
* Recent changes in medication (3 months)
* Current smoking any tobacco use
* Cardiovascular disease, diabetes (Type 1 or 2), and other metabolic or chronic diseases
* More than 7 alcoholic drinks/week of consumption

Ages: 45 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Macrovascular Endothelial function in the fasted condition | 4 weeks
  Endothelial function will be measured via brachial artery flow mediated dilation (ultrasonography) during reactive hyperemia at baseline and after 4 weeks of supplementation.
Microvascular endothelial function in the fasted condition | 4 weeks
  Endothelial function will be measured using forearm muscle oxygenation (near-infrared spectroscopy) will assessed during reactive hyperemia at baseline and after 4 weeks of supplementation.
Microvascular digital endothelial function in the fasted condition | 4 weeks
  Endothelial function will be measured using peripheral (finger) arterial tonometry (EndoPAT device) during reactive hyperemia at baseline and after 4 weeks of supplementation.
Macrovascular Endothelial function during acute hyperglycemia | 4 weeks
  Endothelial function will be measured via brachial artery flow mediated dilation (ultrasonography) during reactive hyperemia at 30, 60, and 90 minutes after oral glucose ingestion at baseline and after 4 weeks of supplementation.
Microvascular forearm endothelial function during acute hyperglycemia | 4 weeks
  Endothelial function will be measured using forearm muscle oxygenation (near-infrared spectroscopy) during reactive hyperemia at 30, 60, and 90 minutes after oral glucose ingestion at baseline and after 4 weeks of supplementation.
Central and peripheral arterial stiffness in the fasted condition | 4 weeks
  Arterial stiffness will be measured using central (carotid-femoral) and peripheral (femoral-ankle) PWV at baseline and after 4 weeks of supplementation.
Central arterial stiffness during acute hyperglycemia | 4 weeks
  Arterial stiffness will be measured using central (carotid-femoral) PWV at 30, 60, and 90 minutes after oral glucose ingestion at baseline and after 4 weeks of supplementation.
Blood pressure in the fasted condition | 4 weeks
  Brachial and aortic blood pressures will be assessed using an automated sphygmomanometry arm cuff (SphygmoCor XCEL). Beat-to-beat blood pressure will be measured using an automated photoplethysmography finger cuff (Fineometer). Blood pressure will be measured at baseline and after 4 weeks of supplementation.
Blood pressure during acute hyperglycemia | 4 weeks
  Brachial and aortic blood pressures (systolic and diastolic) will be assessed using an automated sphygmomanometry arm cuff (SphygmoCor XCEL). Beat-to-beat blood pressure will be measured using an automated photoplethysmography finger cuff (Fineometer). Blood pressure will be measured after an oral glucose ingestion at 30, 60, and 90 minutes at baseline and after 4 weeks of supplementation.
Total peripheral resistance in the fasted condition. | 4 weeks
  Total peripheral resistance will be measured using an automated photoplethysmography finger cuff (Finometer) at baseline and after 4 weeks of supplementation.
Total peripheral resistance during acute hyperglycemia | 4 weeks
  Total peripheral resistance will be measured using an automated photoplethysmography finger cuff (Finometer) at 30, 60, and 90 minutes after oral glucose ingestion at baseline and after 4 weeks of supplementation.
Stroke volume in the fasted condition | 4 weeks
  Stroke volume will be measured using an automated photoplethysmography finger cuff (Finometer) at baseline and after 4 weeks of supplementation.
Stroke volume during acute hyperglycemia | 4 weeks
  Stroke volume will be measured using an automated photoplethysmography finger cuff (Finometer) at 30, 60, and 90 minutes after oral glucose ingestion at baseline and after 4 weeks of supplementation.
24-hour ambulatory blood pressure monitoring | 4 weeks
  An ambulatory blood pressure cuff, measuring blood pressure for 24-hours will be obtained on two separate days at baseline and after 4 weeks of supplementation.

SECONDARY OUTCOMES:
Serum glucose and insulin levels. | 4 weeks
  Serum glucose and insulin levels will be tested at baseline and after 4 weeks of supplementation.
Serum arginine levels | 4 weeks
  Serum L-Arginine levels will be tested at baseline and after 4 weeks of supplementation.
Serum arginase levels | 4 weeks
  Serum arginase levels will be tested at baseline and after 4 weeks of supplementation.
Serum Nitric Oxide levels | 4 weeks
  Serum nitric oxide levels will be tested at baseline and after 4 weeks of supplementation.
Serum Endothelin-1 levels | 4 weeks
  Serum endothelin-1 levels will be tested at baseline and after 4 weeks of supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Figueroa, Principal Investigator — Texas Tech University
Locations (1):
- TTU Kinesiology and Sport Management Building, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maharaj A, Fischer SM, Dillon KN, Kang Y, Martinez MA, Figueroa A. Effects of L-Citrulline Supplementation on Endothelial Function and Blood Pressure in Hypertensive Postmenopausal Women. Nutrients. 2022 Oct 20;14(20):4396. doi: 10.3390/nu14204396. PMID 36297080
- [Background] Figueroa A, Maharaj A, Kang Y, Dillon KN, Martinez MA, Morita M, Nogimura D, Fischer SM. Combined Citrulline and Glutathione Supplementation Improves Endothelial Function and Blood Pressure Reactivity in Postmenopausal Women. Nutrients. 2023 Mar 23;15(7):1557. doi: 10.3390/nu15071557. PMID 37049398
- [Background] Maharaj A, Fischer SM, Dillon KN, Kang Y, Martinez MA, Figueroa A. Acute Citrulline Blunts Aortic Systolic Pressure during Exercise and Sympathoactivation in Hypertensive Postmenopausal Women. Med Sci Sports Exerc. 2022 May 1;54(5):761-768. doi: 10.1249/MSS.0000000000002848. Epub 2022 Jan 3. PMID 34974502
- [Background] McDonald JD, Mah E, Chitchumroonchokchai C, Dey P, Labyk AN, Villamena FA, Volek JS, Bruno RS. Dairy milk proteins attenuate hyperglycemia-induced impairments in vascular endothelial function in adults with prediabetes by limiting increases in glycemia and oxidative stress that reduce nitric oxide bioavailability. J Nutr Biochem. 2019 Jan;63:165-176. doi: 10.1016/j.jnutbio.2018.09.018. Epub 2018 Sep 25. PMID 30412905
- [Background] Figueroa A, Alvarez-Alvarado S, Ormsbee MJ, Madzima TA, Campbell JC, Wong A. Impact of L-citrulline supplementation and whole-body vibration training on arterial stiffness and leg muscle function in obese postmenopausal women with high blood pressure. Exp Gerontol. 2015 Mar;63:35-40. doi: 10.1016/j.exger.2015.01.046. Epub 2015 Jan 28. PMID 25636814